CLINICAL TRIAL: NCT07143539
Title: Early Exercise-based Rehabilitation in High-risk Patients Hospitalized for Acute Pulmonary Embolism: a Pragmatic Multicenter Randomized Partially Blinded Superiority Trial
Brief Title: Early Exercise-Based Rehabilitation in Patients Hospitalized for Acute Pulmonary Embolism
Acronym: RehabPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-01502
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Venous Thromboembolism (VTE); Exercise Therapy; Quality of Life (QOL); Anxiety Depression; Humans; Exercise Tolerance; Rehabilitation Exercise; Dyspnea; Functional Status; Pulmonary Embolism (Diagnosis)
Keywords: pulmonary embolism; deep vein thrombosis; excercise-based rehabilitation; post-PE syndrome; health-related quality of life; anxiety; depression; dyspnea; impact of early excercise-based rehabilitation
MeSH Terms: conditions — Venous Thromboembolism; Dyspnea; Pulmonary Embolism; Disease; Venous Thrombosis; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study staff, blinded to participants' study group allocation, will conduct follow-up visit and assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early exercise-based rehabilitation (EBR) (Active Comparator): Early 6- to 8-week, center-based EBR program, and 2 educational sessions
  Interventions: Other: Exercise-based rehabilitation program
- usual care (no rehabilitation) (No Intervention): Participants in the control group will receive usual care (i.e., no exercise-based rehabilitation program)

INTERVENTIONS:
Other: Exercise-based rehabilitation program — Participants in the intervention group will receive a patient-tailored early (i.e., within 4 weeks of PE diagnosis) EBR program, comprising 16-18 sessions of supervised aerobic exercise and resistance/strength training at local outpatient rehabilitation centers, along with 2 PE-related educational sessions at 2 and 6 weeks of rehabilitation. Participants will receive comprehensive information on the purpose of EBR and each of its components, reassurance on its safety, and education on self-monitoring. Furthermore, physiotherapists will tailor the training based on specific capabilities, focusing on areas of weakness.
  Arms: Early exercise-based rehabilitation (EBR)

SUMMARY:
Up to half of patients with pulmonary embolism (PE) suffer from impaired quality of life, reduced physical capacity, and symptoms like shortness of breath even three months after diagnosis, despite standard treatment with anticoagulation (blood thinners). The randomized RehabPE trial investigates whether an early, structured rehabilitation program with physical training and patient education can prevent such long-term effects.

The study includes hospitalized patients with acute symptomatic PE who are at increased risk of impaired quality of life three months after diagnosis. After informed consent, patients are randomly assigned to one of two groups: one receives an early 6-8-week, center-based rehabilitation program; the other receives standard follow-up care without rehabilitation. The intervention group completes 16-18 outpatient sessions of endurance and strength training, along with two education sessions covering the condition, treatment, and symptom management.

Over 180 days, changes in quality of life, physical exercise capacity, breathlessness, and psychological symptoms, and the time to return to work / usual daily activities will be monitored and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Hospitalization for objectively confirmed acute symptomatic PE, defined as intraluminal filling defect of a segmental or more proximal pulmonary artery on computed tomography pulmonary angiography (CTPA) or a high-probability ventilation-perfusion scintigraphy, and admission within the past 7 days
3. Increased risk for post-PE syndrome, defined as simplified Pulmonary Embolism Severity Index (sPESI) ≥1 point at the time of admission
4. Written informed consent

Exclusion Criteria:

1. Contraindication to EBR (known unstable cardiac conditions like angina pectoris, severe valvular heart disease, or severe resting pulmonary hypertension)
2. Medical condition that clearly precludes participation in EBR (e.g., inability to walk, unstable joints, severe neurological impairment)
3. Recently completed (i.e., <6 months), ongoing, or planned in- or outpatient EBR, or planned supervised outpatient physiotherapy for any indication
4. Planned hospitalization during follow-up (e.g., elective surgery or inpatient chemotherapy)
5. Contraindication to anticoagulation
6. Life expectancy <1 year based on the treating physician's clinical judgement
7. Known pregnancy
8. Inability to speak German or French
9. Participation in another study that prohibits concurrent participation in RehabPE
10. Unable to provide informed consent (e.g., due to dementia)
11. Unwilling to provide informed consent
12. Prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in generic health-related quality of life (Physical Component Summary score; SF-36) | From baseline to day 90 after randomization
  Change from baseline to day 90 after randomization in generic healt-related quality of life (HRQoL) assessed by the PCS score of the self-completed SF-36 questionnaire. The SF-36 consists of 36 questions measuring 8 domains (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health) and assesses generic HRQoL during the previous 30 days. The PCS score is obtained from all 8 domains and ranges from 0 to 100.

SECONDARY OUTCOMES:
Change in generic health-related quality of life (Physical Component Summary score; SF-36) | From baseline to day 180 after randomization
  Change from baseline to day 180 after randomization in the SF-36 Physical Component Summary score, ranging from 0 to 100 with higher scores indicating better HRQoL.
Change in generic health-related quality of life (Mental Component Summary score; SF-36) | From baseline to day 90 and to day 180 after randomization
  Changes from baseline to day 90 and to day 180 after randomization in the SF-36 Mental Component Summary score, ranging from 0 to 100 with higher scores indicating better HRQoL.
Change in PE-specific health-related quality of life (PEmb-QoL) | From baseline to day 90 and to day 180 after randomization
  Change from baseline to day 90 and to day 180 after randomization in PE-specific health-realted quality of life assessed by the self-completed PEmb-QoL questionnaire, which comprises 9 questions covering 6 domains, with scores ranging from 0 to 100. Total scores will be calculated based on the average of scores of all 6 domains.
Change in physical exercise capacity (6 minute walking test) | From baseline to day 90 and to day 180 after randomization
  Change in physical exercise capacity from baseline to day 90 and to day 180 after randomization will be measured by the 6 minute walking test (6MWT). Participants will be asked to walk as far as possible in 6 minutes along a flat corridor of at least 30 mesters under supervision, and the distance in meters will determine the 6MWD.
Change in functional status (Post-VTE Functional Status) | From baseline to day 90 and to day 180 after randomization
  Change in functional status will be assessed by the Post-VTE Functional Status scale, where patients will grade their functional status on a scale ranging from 0 (no limitations due to VTE symptoms) to 4 (depending on assistance in activities of daily living due to VTE symptoms).
Time to return to work (workers) or usual activities of daily living (non-workers) | For the duration of the study: 180 days
  Time (days) to return to work in workers or to usual activities of daily living in non-workers will be obtained based on information from patient interviews.
Change in dyspnea | From baseline to day 90 and to day 180 after randomization
  Dyspnea will be measured based on information from patient interviews, using the NYHA classification, ranging from 1 (no limitation of physical activity due to shortness of breath) to 4 (unable to carry on any physical activity without shortness of breath).
Change in symptoms of anxiety (GAD-7) | From baseline to day 90 and to day 180 after randomization
  Change in symptoms of anxiety will be assessed by the self-completed General Anxiety Disorder 7 (GAD-7) ranging from 0 to 21 points.
Change in symptoms of depression (PHQ-9) | From baseline to day 90 and to day 180 after randomization
  Change in symptoms of depression will be assessed by the self-completed Patient Health Questionnaire 9 (PHQ-9), ranging from 0 to 27 points.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Tritschler, MD, MSc, Principal Investigator — Inselspital, Universitätsspital Bern
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After publication of the study results, an anonymized data set relating to the primary publication along with the latest version of the study protocol, the informed consent form, the statistical analysis plan, and the code used for the analyses will be made publicly available for replication of the study results and secondary data analyses (upon request) in the Bern Open Repository and Information System (BORIS) Research Data, an online non-commercial data repository that meets Swiss National Science Foundation requirements for FAIR Data Principles (www.force11.org/group/fairgroup/fairprinciples)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After publication of the study results
Access Criteria: Data will be publicly available for replication of the study results and secondary data analyses (upon request) in the Bern Open Repository and Information System (BORIS) Research Data.
URL: https://boris-portal.unibe.ch/

REFERENCES:
- [Background] Luijten D, de Jong CMM, Ninaber MK, Spruit MA, Huisman MV, Klok FA. Post-Pulmonary Embolism Syndrome and Functional Outcomes after Acute Pulmonary Embolism. Semin Thromb Hemost. 2023 Nov;49(8):848-860. doi: 10.1055/s-0042-1749659. Epub 2022 Jul 12. PMID 35820428
- [Background] Keller K, Tesche C, Gerhold-Ay A, Nickels S, Klok FA, Rappold L, Hasenfuss G, Dellas C, Konstantinides SV, Lankeit M. Quality of life and functional limitations after pulmonary embolism and its prognostic relevance. J Thromb Haemost. 2019 Nov;17(11):1923-1934. doi: 10.1111/jth.14589. Epub 2019 Aug 13. PMID 31344319
- [Background] Sista AK, Klok FA. Late outcomes of pulmonary embolism: The post-PE syndrome. Thromb Res. 2018 Apr;164:157-162. doi: 10.1016/j.thromres.2017.06.017. Epub 2017 Jun 16. PMID 28641836
- [Background] Yu A, Ding W, Lin W, Cai J, Huang W. Application of pulmonary rehabilitation in patients with pulmonary embolism (Review). Exp Ther Med. 2022 Jan;23(1):96. doi: 10.3892/etm.2021.11019. Epub 2021 Dec 1. PMID 34976138
- [Background] Cires-Drouet RS, Mayorga-Carlin M, Toursavadkohi S, White R, Redding E, Durham F, Dondero K, Prior SJ, Sorkin JD, Lal BK. Safety of exercise therapy after acute pulmonary embolism. Phlebology. 2020 Dec;35(10):824-832. doi: 10.1177/0268355520946625. Epub 2020 Jul 27. PMID 32720853
- [Background] Amoury M, Noack F, Kleeberg K, Stoevesandt D, Lehnigk B, Bethge S, Heinze V, Schlitt A. Prognosis of patients with pulmonary embolism after rehabilitation. Vasc Health Risk Manag. 2018 Aug 30;14:183-187. doi: 10.2147/VHRM.S158815. eCollection 2018. PMID 30214219
- [Background] Gleditsch J, Jervan O, Haukeland-Parker S, Tavoly M, Geier O, Holst R, Klok FA, Johannessen HH, Ghanima W, Hopp E. Effects of pulmonary rehabilitation on cardiac magnetic resonance parameters in patients with persistent dyspnea following pulmonary embolism. Int J Cardiol Heart Vasc. 2022 Mar 23;40:100995. doi: 10.1016/j.ijcha.2022.100995. eCollection 2022 Jun. PMID 35345773
- [Background] Albaghdadi MS, Dudzinski DM, Giordano N, Kabrhel C, Ghoshhajra B, Jaff MR, Weinberg I, Baggish A. Cardiopulmonary Exercise Testing in Patients Following Massive and Submassive Pulmonary Embolism. J Am Heart Assoc. 2018 Mar 3;7(5):e006841. doi: 10.1161/JAHA.117.006841. PMID 29502109
- [Background] Rolving N, Brocki BC, Bloch-Nielsen JR, Larsen TB, Jensen FL, Mikkelsen HR, Ravn P, Frost L. Effect of a Physiotherapist-Guided Home-Based Exercise Intervention on Physical Capacity and Patient-Reported Outcomes Among Patients With Acute Pulmonary Embolism: A Randomized Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e200064. doi: 10.1001/jamanetworkopen.2020.0064. PMID 32108888
- [Background] Ghram A, Jenab Y, Soori R, Choobineh S, Hosseinsabet A, Niyazi S, Shirani S, Shafiee A, Jalali A, Lavie CJ, Wisloff U. High-Intensity Interval Training in Patients with Pulmonary Embolism: A Randomized Controlled Trial. Med Sci Sports Exerc. 2021 Oct 1;53(10):2037-2044. doi: 10.1249/MSS.0000000000002680. PMID 33867496
- [Background] Lakoski SG, Savage PD, Berkman AM, Penalosa L, Crocker A, Ades PA, Kahn SR, Cushman M. The safety and efficacy of early-initiation exercise training after acute venous thromboembolism: a randomized clinical trial. J Thromb Haemost. 2015 Jul;13(7):1238-44. doi: 10.1111/jth.12989. Epub 2015 May 25. PMID 25912176
- [Background] Jervan O, Haukeland-Parker S, Gleditsch J, Tavoly M, Klok FA, Steine K, Johannessen HH, Spruit MA, Atar D, Holst R, Astrup Dahm AE, Sirnes PA, Stavem K, Ghanima W. The Effects of Exercise Training in Patients With Persistent Dyspnea Following Pulmonary Embolism: A Randomized Controlled Trial. Chest. 2023 Oct;164(4):981-991. doi: 10.1016/j.chest.2023.04.042. Epub 2023 May 5. PMID 37149257
- [Background] Boon GJAM, Janssen SMJ, Barco S, Bogaard HJ, Ghanima W, Kroft LJM, Meijboom LJ, Ninaber MK, Nossent EJ, Spruit MA, Symersky P, Vliegen HW, Vonk Noordegraaf A, Huisman MV, Siegerink B, Abbink JJ, Klok FA. Efficacy and safety of a 12-week outpatient pulmonary rehabilitation program in Post-PE Syndrome. Thromb Res. 2021 Oct;206:66-75. doi: 10.1016/j.thromres.2021.08.012. Epub 2021 Aug 17. PMID 34419865
- [Background] van Es J, den Exter PL, Kaptein AA, Andela CD, Erkens PM, Klok FA, Douma RA, Mos IC, Cohn DM, Kamphuisen PW, Huisman MV, Middeldorp S. Quality of life after pulmonary embolism as assessed with SF-36 and PEmb-QoL. Thromb Res. 2013 Nov;132(5):500-5. doi: 10.1016/j.thromres.2013.06.016. Epub 2013 Oct 3. PMID 24090607
- [Background] Kahn SR, Akaberi A, Granton JT, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Hernandez P, Aaron SD, Hirsch AM. Quality of Life, Dyspnea, and Functional Exercise Capacity Following a First Episode of Pulmonary Embolism: Results of the ELOPE Cohort Study. Am J Med. 2017 Aug;130(8):990.e9-990.e21. doi: 10.1016/j.amjmed.2017.03.033. Epub 2017 Apr 8. PMID 28400247
- [Background] Kahn SR, Hirsch AM, Akaberi A, Hernandez P, Anderson DR, Wells PS, Rodger MA, Solymoss S, Kovacs MJ, Rudski L, Shimony A, Dennie C, Rush C, Geerts WH, Aaron SD, Granton JT. Functional and Exercise Limitations After a First Episode of Pulmonary Embolism: Results of the ELOPE Prospective Cohort Study. Chest. 2017 May;151(5):1058-1068. doi: 10.1016/j.chest.2016.11.030. Epub 2016 Dec 6. PMID 27932051
- [Background] Klok FA, van Kralingen KW, van Dijk AP, Heyning FH, Vliegen HW, Huisman MV. Prevalence and potential determinants of exertional dyspnea after acute pulmonary embolism. Respir Med. 2010 Nov;104(11):1744-9. doi: 10.1016/j.rmed.2010.06.006. PMID 20599368
- [Background] Klok FA, Ageno W, Ay C, Back M, Barco S, Bertoletti L, Becattini C, Carlsen J, Delcroix M, van Es N, Huisman MV, Jara-Palomares L, Konstantinides S, Lang I, Meyer G, Ni Ainle F, Rosenkranz S, Pruszczyk P. Optimal follow-up after acute pulmonary embolism: a position paper of the European Society of Cardiology Working Group on Pulmonary Circulation and Right Ventricular Function, in collaboration with the European Society of Cardiology Working Group on Atherosclerosis and Vascular Biology, endorsed by the European Respiratory Society. Eur Heart J. 2022 Jan 25;43(3):183-189. doi: 10.1093/eurheartj/ehab816. PMID 34875048
- [Background] Boon GJAM, Huisman MV, Klok FA. Determinants and Management of the Post-Pulmonary Embolism Syndrome. Semin Respir Crit Care Med. 2021 Apr;42(2):299-307. doi: 10.1055/s-0041-1722964. Epub 2021 Feb 6. PMID 33548930
- [Background] Sista AK, Miller LE, Kahn SR, Kline JA. Persistent right ventricular dysfunction, functional capacity limitation, exercise intolerance, and quality of life impairment following pulmonary embolism: Systematic review with meta-analysis. Vasc Med. 2017 Feb;22(1):37-43. doi: 10.1177/1358863X16670250. Epub 2016 Oct 5. PMID 27707980